CLINICAL TRIAL: NCT01285011
Title: Short Term Follow-up of Patient Implanted With the Proximal Interphalangeal
Brief Title: Short Term Follow-up of Patient Implanted With the Proximal Interphalangeal Implant
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Services (Industry)
Responsible Party: Sponsor
Other Study IDs: RECON-EMEA-08
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Hammer Toe; Claw Toe; Shortening 2nd Toe; Revision of Arthrodesis or Arthroplasty Failure
Keywords: arthrodesis; PIP joint
MeSH Terms: conditions — Hammer Toe Syndrome; Ankylosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ipp-On: Patient implanted with the Ipp-On

SUMMARY:
Hammertoe and ClawToe are ones of the most common foot deformities. The second toe is the most frequently affected, but the other small toes may also be involved. When nonoperative treatment fails, surgery often is recommended. One surgical option is the arthrodesis of the Proximal Interphalangeal (PIP) joint. This arthrodesis is technically demanding, its needs:

* Internal fixation;
* Interphalangeal Compression;
* Anatomic PIP joint plantar flexion angle. The implant Ipp-On has been developed for this specific arthrodesis. The objective of this study is to evaluate the efficacy and safety of the Proximal Interphalangeal Implant: Ipp-On at short term follow up.

The safety of the Ipp-On will be described in terms of rate of device related complications.

The efficacy of the Ipp-On will be described in terms of fusion rate at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who needs a proximal interphalangeal joint arthrodesis for whose surgeon has recommended that a proximal Interphalangeal Implant Ipp-On be implanted
* Age >= 18 years
* Have willingness to give his/her Data Transfer Authorization

Exclusion Criteria:

* Contraindication of the implantation of the Ipp-On The implant should not be used in a patient who has currently, or who has a history of: • Active local or systemic infection

  * Severe peripheral vascular disease
  * Severe longitudinal deformity
  * Insufficient quantity or quality of bone to permit stabilization of the arthrodesis
  * Conditions that restrict the patient's ability or willingness to follow postoperative instructions during the healing process
  * Suspected or documented metal allergy or intolerance.
* History of prior mental illness or patient demonstrates that their mental capacity may interfere with their ability to follow the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient who needs a proximal interphalangeal joint arthrodesis for whose surgeon has recommended that a proximal Interphalangeal Implant Ipp-On be implanted
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2009-04; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Rate of device related complications | 12 months
fusion rate | 6 months

SECONDARY OUTCOMES:
Fusion rate | 3 months
American Orthopaedic Foot and Ankle Society Lesser Metatarsophalangeal Scale (AOFAS LMIS) score | 6 months/12 months
Radiological Evaluation | 6 months/12 months
Clinical Assessment | 6 months/12 months
Subjective assessment | 6 months/12 months

CONTACTS AND LOCATIONS:
Locations (5):
- Sint Lucas Clinic, Bruges, Belgium
- France (3):
  - CHU Pellegrin, Bordeaux
  - Clinique du Parc, Lyon
  - ICP, Paris
- Ospedale Regionale di Bellinzona e Valli, Bellinzona, Switzerland